CLINICAL TRIAL: NCT01372215
Title: Multi-Compression Spot Mammography
Status: Terminated | Type: Observational
Why Stopped: Referral physician no longer available
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Kent Ogden, PhD, State University of New York - Upstate Medical University
Other Study IDs: SUNYUMU 5907
Record Dates: First submitted 2011-06-10; First posted 2011-06-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Breast Diseases
Keywords: Breast mass; Breast lesion
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study, participants, who are scheduled to have a breast biopsy, will have several extra spot mammogram images taken of the suspicious area. These images will be acquired with varying levels of compression. The images will then be analyzed to determine whether the type of lesion (malignant or benign) can be determined from the image data alone. The biopsy results will be used as a gold standard to determine the true malignancy status

ELIGIBILITY:
Inclusion Criteria:

* Women 45 years and older
* Women with suspicious mammography findings requiring a biopsy

Exclusion Criteria:

* Men
* Pregnant women

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women 45 years of age and older who have a suspicious mammagraphy requiring a biopsy
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2011-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kent Ogden, PhD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- University Health Care Center (UHCC), Syracuse, New York, United States